CLINICAL TRIAL: NCT02660762
Title: A Prospective Phase II Trial of Modified MRC UKALL Ⅻ/ECOG E2993 Regimen in the Treatment of Low Risk Philadelphia Chromosome Negative Acute Lymphoblastic Leukemia for Young Adults
Brief Title: Modified MRCUKALLⅫ/ECOGE2993 Regimen for ALL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, dr. luyue, professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-ALL-5010
Record Dates: First submitted 2016-01-13; First posted 2016-01-21 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Leukaemia,Lymphoblastic
MeSH Terms: conditions — Leukemia | interventions — Vincristine; Daunorubicin; pegaspargase; Prednisone; Methotrexate; Cyclophosphamide; Cytarabine; Mercaptopurine; Etoposide; Dexamethasone; Thioguanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Modified MRCUKALLⅫ/ECOGE2993 Regimen (Experimental): All patients received phase 1 of induction therapy, which consisted of daunorubicin,vincristine,Pegaspargase,prednisone and methotrexate (intrathecally).Patients went on to phase 2 at the end of phase 1.Phase 2 therapy consisted of cyclophosphamide,cytarabine,6-Mercaptopurine and methotrexate intrathecally. After Induction therapy, all patients received intensification therapy with high-dose methotrexate followed by Pegaspargase. After intensification therapy,patients received consolidation(cytarabine, etoposide,Pegaspargase,dexamethasone,vincristine,cyclophosphamide,daunorubicin,thioguanine)and maintenance therapy(vincristine,6-mercaptopurine,methotrexate
  ,prednisone). Intrathecal methotrexate and intrathecal cytarabine were given as CNS prophylaxis.
  Interventions: Drug: Vincristine; Drug: Daunorubicin; Drug: Pegaspargase; Drug: Prednisone; Drug: Intrathecal Methotrexate; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: 6-Mercaptopurine; Drug: Methotrexate; Drug: Etoposide; Drug: dexamethasone; Drug: thioguanine; Drug: intrathecal cytarabine

INTERVENTIONS:
Drug: Vincristine — induction therapy I：1.4 mg/m2 IV d1, 8, 15, 22； consolidation therapy(Cycle 1)：1.4 mg/m2 IV d1, 8, 15, 22； Maintenance therapy: 1.4 mg/m2 intravenously every 3 months for a total of 2.5 years
  Other Names: Vincasar
Drug: Daunorubicin — induction therapy I：60 mg/m2 IV d1, 8, 15, 22； consolidation therapy(Cycle 3)：25 mg/m2 IV d1, 8, 15, 22；
  Other Names: Cerubidine
Drug: Pegaspargase — induction therapy I: 2500U/m2,im,d8,22 Intensification therapy:2500U/m2 im, d2,23 consolidation therapy(Cycle 2，4)：2500U/m2 im, d1
  Other Names: Oncaspar
Drug: Prednisone — induction therapy I：60 mg/m2 PO d1-28; Maintenance therapy:prednisone 60 mg/m2 orally for 5 days every 3 months for a total of 2.5 years
  Other Names: Prednisone acetate
Drug: Intrathecal Methotrexate — induction therapy I：12.5 mg IT d15 induction therapy II：12.5 mg IT d1, 8, 15, 22
  Other Names: Rheumatrex
Drug: Cyclophosphamide — induction therapy II:650 mg/m2 IV d1, 15, 29 consolidation therapy(Cycle 3)：650 mg/m2 IV，d29
  Other Names: Cytoxan
Drug: Cytarabine — induction therapy II:75 mg/m2 IV d1-4, 8-11, 15-18, 22-25 consolidation therapy(Cycle 1，2，4)：75 mg/m2 intravenously on days 1 to 5 consolidation therapy(Cycle 3):75 mg/m2 intravenously on days 31 to 34 and 38 to 41
  Other Names: Cytosar-U
Drug: 6-Mercaptopurine — induction therapy II:60 mg/m2 PO d1-28 Maintenance therapy:75 mg/m2 orally each day for a total of 2.5 years
  Other Names: Purinethol
Drug: Methotrexate — Intensification therapy:3 g/m2 intravenously given on days 1, 8, and 22 Maintenance therapy:20 mg/m2 orally or intravenously once a week for a total of 2.5 years.
  Other Names: Rheumatrex
Drug: Etoposide — consolidation therapy(Cycle 1，2，4)：100 mg/m2 intravenously on days 1 to 5
  Other Names: VePesid
Drug: dexamethasone — consolidation therapy(Cycle 1)：10mg/m2 orally on days 1 to 28
  Other Names: Dexamethasone Sodium
Drug: thioguanine — consolidation therapy(Cycle 3): 60 mg/m2 orally on days 29 to 42
  Other Names: 6-TG
Drug: intrathecal cytarabine — 50 mg intrathecal cytarabine was given on 4 occasions 3 months apart during maintenance therapy.
  Other Names: Cytosar-U

SUMMARY:
This prospective study was conducted to evaluate the efficacy and safety profiles of Modified MRCUKALLⅫ/ECOGE2993 Regimen in young adults with newly diagnosed, low-risk, Philadelphia chromosome negative acute lymphoblastic leukaemia.

DETAILED DESCRIPTION:
All patients received a modified BFM regimen which was derived from the MRCUKALLⅫ/ECOGE2993 Regimen.The differences were as follows:(1) cranial prophylactic radiotherapy was omitted (2) Pegaspargase was used instead of L- asparaginase for patient.(3)Two additional Pegaspargase treatments were added into consolidation therapy.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed ALL
* age:18-35years
* WBC count below 30×109/L(B lineage)；WBC count below 100×109/L(T lineage)
* absence of t(9;22), t(1;19), t(4;11) or any other 11q23 rearrangements
* receive no chemotherapy or radiotherapy before
* Adequate renal function (eg, serum creatinine≤1.5 mg/dL and creatinine clearance ≥50 mL minute), and hepatic function (e.g, total bilirubin≤ 2 times the upper limit of normal and aspartate and alanine transaminase levels ≤ 3 times the upper limit of normal)

Exclusion Criteria:

* mismatch the inclusion criteria
* systematic central nervous system involvement, previous or concomitant malignancies and any coexisting medical problems that could cause poor compliance with the study protocol.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
progression free survival | up to end of follow-up-phase (approximately 3 years)

SECONDARY OUTCOMES:
overall survival | up to end of follow-up-phase (approximately 3 years)
complete remission rate | every 4 weeks,up to completion of induction treatment(approximately 2months)
Incidence of Treatment-Emergent Adverse Events classified according to Common Terminology Criteria for Adverse Events v3.0 (CTCAE) | up to end of follow-up-phase (approximately 3 years)
  including hematological safety and non-hematological safety.
Minimal Residual Disease (MRD) monitoring | During treatment at time point 4, 8, 12, 16,20,24, 28 weeks（every 4 weeks,up to completion of consolidation therapy）and 40，52，64，76，88，100，112，124 weeks( every 12 weeks during maintenance therapy,up to the end of treatment )
  Minimal residual disease is measured in bone marrow using an multiparameter flow cytometry.For the patients who achieved complete remission after induction therapy, if two consecutive tests for MRD were positive,we will define it as MRD positive

CONTACTS AND LOCATIONS:
Overall Officials: yue lu, MD., Principal Investigator — Department of Hematological Oncology, Sun Yat-sen University Cancer Center; State Key Laboratory of Oncology in South China
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Rowe JM, Buck G, Burnett AK, Chopra R, Wiernik PH, Richards SM, Lazarus HM, Franklin IM, Litzow MR, Ciobanu N, Prentice HG, Durrant J, Tallman MS, Goldstone AH; ECOG; MRC/NCRI Adult Leukemia Working Party. Induction therapy for adults with acute lymphoblastic leukemia: results of more than 1500 patients from the international ALL trial: MRC UKALL XII/ECOG E2993. Blood. 2005 Dec 1;106(12):3760-7. doi: 10.1182/blood-2005-04-1623. Epub 2005 Aug 16. PMID 16105981